CLINICAL TRIAL: NCT02748434
Title: Glucose Variability in Subclinical Hypertrophy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Graydon Meneilly, Professor, UBC Department of Medicine, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: H16-01025
Record Dates: First submitted 2016-04-20; First posted 2016-04-22 (Estimated); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Mellitus; Lipohypertrophy
Keywords: iPro2 Continuous Blood Glucose Recorder; Subclinical
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lipohypertrophy (Other): Participants inject their insulin into the abdomen into areas of lipohypertrophy that were identified by ultrasound in Phase 1 of the study.
  Interventions: Other: Lipohypertrophy
- Normal Subcutaneous Tissue (Other): Participants inject their insulin into the abdomen into areas with normal subcutaneous tissue.
  Interventions: Other: Normal Subcutaneous Tissue

INTERVENTIONS:
Other: Lipohypertrophy
  Arms: Lipohypertrophy
Other: Normal Subcutaneous Tissue
  Arms: Normal Subcutaneous Tissue

SUMMARY:
Evaluation of insulin absorption at sites affected by clinically apparent lipohypertrophy through short-term continuous glucose monitoring has shown inconsistent results and it is yet unknown how or if subclinical lipohypertrophy affects absorption. In this study investigators propose to enroll at least 20 people who participated in phase 1 and who were determined to have subclinical lipohypertrophy to examine the correlation between glycemic control and amount of insulin injected in subclinical hypertrophic areas using capillary blood glucose and continuous glucose monitoring.

DETAILED DESCRIPTION:
Patients will be randomized and data interpreters will be blinded to two alternating six-day protocols where the patients will be advised verbally and by written instruction to inject insulin in sites of subclinical lipohypertrophy or normal subcutaneous tissue. Patients will be asked to monitor and record their capillary blood glucose with meals and prior to bedtime using their own capillary blood glucose monitor. A trained research nurse at the Diabetes Centre will instrument each patient with an iPro 2 glucose sensor (Medtronic Canada). These sensors continuously measure blood glucose for periods of up to 7 days. A trained nurse will clean the skin with a superficial disinfectant and a small catheter will be inserted in the subcutaneous tissue at a non-lipohypertrophic site. The catheter will then be attached to a glucose sensor. Patients will wear this sensor for two periods of 6 days each at different sites. At the end of each of the two six day periods, the sensor will be removed.

ELIGIBILITY:
Inclusion Criteria:

* Participation in phase 1
* Type 1 or Type 2 diabetes for at least 2 years
* Using insulin to manage diabetes
* At least 19 years of age

Exclusion Criteria:

* Taking insulin secretagogues (gliclazide, glyburide, glipizide
* Taking other injectable diabetes medications (i.e. liraglutide, Victoza)
* Taking systemic steroids (e.g. prednisone)
* Not fluent in speaking and writing English (unless accompanied by a translator)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Blood glucose levels | Continuously for 12 days
  iPro2 Continuous Blood Glucose Monitor

CONTACTS AND LOCATIONS:
Overall Officials: Graydon Meneilly, MD, Principal Investigator — University of British Columbia; Jordanna Kapeluto, MD, Principal Investigator — University of British Columbia; Breay Paty, MD, Principal Investigator — University of British Columbia
Locations (2):
- Canada (2):
  - Gerontology Research Lab, Vancouver, British Columbia
  - Vancouver General Hospital Diabetes Centre, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: No